CLINICAL TRIAL: NCT05571462
Title: Mobility and Activity Patterns in Hospitalised Patients With Severe Acquired Brain Injury Undergoing Rehabilitation. The MAP-study.
Brief Title: Mobility and Activity Patterns in Hospitalised Severe Brain Injury
Acronym: MAP-ABI
Status: Active, not recruiting | Type: Observational
Sponsor: Christian Riberholt (Other)
Collaborators: SENS Innovation Aps (Unknown)
Responsible Party: Sponsor-Investigator, Christian Riberholt, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-22031667
Record Dates: First submitted 2022-09-29; First posted 2022-10-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Brain Injuries
Keywords: Exercise; Physical activity
MeSH Terms: conditions — Brain Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Activity monitor group: No intervention will be applied. All patients will have activity monitors placed at the distal part of the femur and on the torso. Normal rehabilitation will be performed as usual.
  Interventions: Other: Activity monitor group

INTERVENTIONS:
Other: Activity monitor group — No intervention will be applied. All included patients will be monitored with body-worn physical activity monitors during two periods.

SUMMARY:
The purpose of this observational study is to quantify physical activity patterns in patients with severe acquired brain injury admitted for in-hospital rehabilitation.

DETAILED DESCRIPTION:
Patients admitted for rehabilitation will be included for two periods of one-week monitorization of physical activity. The investigators will include all patients with moderate to severe brain injury.

This is an observational cross-sectional study including patients 18 years or above. Patients with conditions such as unstable fractures that restricts mobilisation are excluded. Physical activity is measured continuously during rehabilitation at two separate seven-day periods using a body-worn activity tracker. The first period will be initiated in the early phase of rehabilitation (3 days after admission) and the second at the late phase (10 days before discharge).

Baseline variables considered predictors, confounders or modifiers for physical activity will be collected along with registration of variables during the measurement periods and functional outcome variables at discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old

Exclusion Criteria:

* Planned discharge within two weeks
* Fractures of lower extremities, pelvis or spine prohibiting weight-bearing
* Amputation of lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired brain injury of any cause admitted for rehabilitation at the department will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Early physical activity | Continuous measure of physical activity during day three to ten of rehabilitation
  Activity data collected in the early phase will be the exposure variable. Amount of minutes patients are physically active.

SECONDARY OUTCOMES:
Late physical activity | Continuous measure of physical activity during day three to ten before discharge from rehabilitation
  Activity data collected in the early phase will be the exposure variable. Amount of minutes patients are physically active.
Functional Independence Measure (discharge) | Discharge from rehabilitation (3 months)
  Functional scale evaluating independence from a score of 18 (worst) to 126 (best)
Glasgow Coma Scale (GCS) (admission) | Admission
  Coma scale with score between 3 (worst) to 15 (best)
Comorbidities at admission | Admission
  Number of comorbidities
Early Functional Ability (EFA) score | Admission
  Early signs of functional ability. Score between 20 (worst) and 100 (best)
Ranchos Los Amigos Score | Admission
  Level of cognitive function. Score between 1 (worst) and 8 (best)
Length of stay at intensive care unit | Retrospectively recorded at admission to the rehabilitation department
  Number of days at intensive care unit before admission to rehabilitation unit
Agitated Behaviour Scale (ABS) | Day three to ten of rehabilitation
  Days with ABS above 22. Dichotomised outcome with scores above 22 indicating agitated behaviour.

OTHER OUTCOMES:
Complications during rehabilitation | Rehabilitation period (3 months)
  Registration of the number of complications during rehabilitation stay at hospital (e.g. pneumonia, unrinary infection, hydrocephalus etc). Predefined in protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Wagner, MsC, Principal Investigator — Rigshospitalet, Department of Brain and Spinal Cord Injury
Locations (1):
- Department of Brain and Spinal Cord Injury, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data that are truly anonymised will be uploaded to Zenodo after the publication of the study. Data that we are not able to truly anonymise will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Two years after study completion. Data will be available for at least ten years.
Access Criteria: Any researcher can make contact to primary investigator or sponsor with pre-planned project description.

REFERENCES:
- [Background] Okely AD, Kontsevaya A, Ng J, Abdeta C. 2020 WHO guidelines on physical activity and sedentary behavior. Sports Med Health Sci. 2021 May 14;3(2):115-118. doi: 10.1016/j.smhs.2021.05.001. eCollection 2021 Jun. PMID 35782159
- [Background] Zeiler SR, Krakauer JW. The interaction between training and plasticity in the poststroke brain. Curr Opin Neurol. 2013 Dec;26(6):609-16. doi: 10.1097/WCO.0000000000000025. PMID 24136129
- [Background] Nielsen JB, Willerslev-Olsen M, Christiansen L, Lundbye-Jensen J, Lorentzen J. Science-based neurorehabilitation: recommendations for neurorehabilitation from basic science. J Mot Behav. 2015;47(1):7-17. doi: 10.1080/00222895.2014.931273. PMID 25575219
- [Background] Larsen RT, Wagner V, Korfitsen CB, Keller C, Juhl CB, Langberg H, Christensen J. Effectiveness of physical activity monitors in adults: systematic review and meta-analysis. BMJ. 2022 Jan 26;376:e068047. doi: 10.1136/bmj-2021-068047. PMID 35082116
- [Background] Ferguson T, Olds T, Curtis R, Blake H, Crozier AJ, Dankiw K, Dumuid D, Kasai D, O'Connor E, Virgara R, Maher C. Effectiveness of wearable activity trackers to increase physical activity and improve health: a systematic review of systematic reviews and meta-analyses. Lancet Digit Health. 2022 Aug;4(8):e615-e626. doi: 10.1016/S2589-7500(22)00111-X. PMID 35868813
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. Epidemiology. 2007 Nov;18(6):805-35. doi: 10.1097/EDE.0b013e3181577511. PMID 18049195
- [Background] Pedersen BS, Kristensen MT, Josefsen CO, Lykkegaard KL, Jonsson LR, Pedersen MM. Validation of Two Activity Monitors in Slow and Fast Walking Hospitalized Patients. Rehabil Res Pract. 2022 May 16;2022:9230081. doi: 10.1155/2022/9230081. eCollection 2022. PMID 35615755
- [Background] Riberholt CG, Wagner V, Lindschou J, Gluud C, Mehlsen J, Moller K. Early head-up mobilisation versus standard care for patients with severe acquired brain injury: A systematic review with meta-analysis and Trial Sequential Analysis. PLoS One. 2020 Aug 13;15(8):e0237136. doi: 10.1371/journal.pone.0237136. eCollection 2020. PMID 32790771
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Kramer SF, Hung SH, Brodtmann A. The Impact of Physical Activity Before and After Stroke on Stroke Risk and Recovery: a Narrative Review. Curr Neurol Neurosci Rep. 2019 Apr 22;19(6):28. doi: 10.1007/s11910-019-0949-4. PMID 31011851
- [Background] Fini NA, Bernhardt J, Said CM, Billinger SA. How to Address Physical Activity Participation After Stroke in Research and Clinical Practice. Stroke. 2021 Jun;52(6):e274-e277. doi: 10.1161/STROKEAHA.121.034557. Epub 2021 May 6. No abstract available. PMID 33951930
- [Result] Adey-Wakeling Z, Jolliffe L, O'Shannessy E, Hunter P, Morarty J, Cameron ID, Liu E, Lannin NA. Activity, Participation, and Goal Awareness After Acquired Brain Injury: A Prospective Observational Study of Inpatient Rehabilitation. Ann Rehabil Med. 2021 Dec;45(6):413-421. doi: 10.5535/arm.21034. Epub 2021 Dec 31. PMID 35000366
- [Result] Norvang OP, Hokstad A, Taraldsen K, Tan X, Lydersen S, Indredavik B, Askim T. Correction to: Time spent lying, sitting, and upright during hospitalization after stroke: a prospective observation study. BMC Neurol. 2019 Jan 11;19(1):8. doi: 10.1186/s12883-018-1226-x. PMID 30634934
- [Result] Kjeldsen SS, Brodal L, Brunner I. Activity and rest in patients with severe acquired brain injury: an observational study. Disabil Rehabil. 2022 Jun;44(12):2744-2751. doi: 10.1080/09638288.2020.1844317. Epub 2020 Nov 8. PMID 33161752
- [Derived] Wagner V, Gravesen P, Ghaziani E, Olsen MH, Riberholt CG. Mapping physical activity patterns in hospitalised patients with moderate to severe acquired brain injury - MAP-ABI: Protocol for an observational study. Heliyon. 2023 Nov 8;9(11):e21927. doi: 10.1016/j.heliyon.2023.e21927. eCollection 2023 Nov. PMID 38034693
- See also: Wagner V, Gravesen P, Ghaziani E, Olsen MH, Riberholt CG. Mapping physical activity patterns in hospitalised patients with moderate to severe acquired brain injury - MAP-ABI: Protocol for an observational study. Heliyon. 2023 Nov 8;9(11):e21927. — https://doi.org/10.1016/j.heliyon.2023.e21927